CLINICAL TRIAL: NCT05647291
Title: Pain Relief and Functional Improvement Provided by ESWT in Plantar Fasciitis is Better Than Corticosteroid Injection and Kinesiotherapy: A Randomized Trial
Brief Title: Is ESWT Better in Plantar Fasciitis Treatment?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Collaborators: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ozlem Orhan, Assistant prof, Harran University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HRU/21.17.30
Record Dates: First submitted 2022-11-23; First posted 2022-12-12 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Plantar Fascitis
Keywords: ESWT; Kinesiotaping; corticosteroid injection
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- extracorporeal Shock wave therapy (ESWT) (Experimental): ESWT was performed by the same physician. The applicator was placed at the point of maximum sensitivity. Two thousand pulses with a frequency of 6 Hz and a pressure of 3 bar were applied to patients with an Auto Wave 695 (Mettler electronics, USA) brand device. Patients underwent two sessions of ESWT per week for two weeks, adding up to a total of 4 sessions. Local or regional anesthesia was not administered to any patient during ESWT.
  Interventions: Device: extracorporeal Shock wave therapy
- Kinesiotaping (Active Comparator): Kinesio tape (KinesioTex, KinesioTaping, US) was applied to the relevant extremity of the patient by the physical therapy and rehabilitation physician once a week, three times in total. During KT, the patient was positioned with the knee and ankle joints in the neutral position. The first strip was adhered along the plantar fascia from the calcaneus to the toes using maximum stretch. The other four strips of tape were attached medially and laterally to support the medial longitudinal arch with a 45° inclination. While maximum stretching was applied to the middle 1/3 of all bands, no stretching was applied to the ends.
  Interventions: Device: Kinesiotaping
- Corticosteroid injection (Active Comparator): In the CI group, 40mg/1ml methylprednisolone was applied from the inferior-medial side of the heel to the most sensitive area of the calcaneus medial tubercle of the plantar fascia. The same physician performed a total of two sessions once a week.
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Device: extracorporeal Shock wave therapy — Two thousand pulses with a frequency of 6 Hz and a pressure of 3 bar were applied to patients with an Auto Wave 695 (Mettler electronics, USA) brand device. Patients underwent two sessions of ESWT per week, for two weeks, adding up to a total of 4 sessions.
  Other Names: an Auto Wave 695 (Mettler electronics, USA) brand device
  Arms: extracorporeal Shock wave therapy (ESWT)
Drug: Corticosteroid injection — 40mg/1ml methylprednisolone, two sessions once a week
  Other Names: methylprednisolone
  Arms: Corticosteroid injection
Device: Kinesiotaping — The first strip was adhered along the plantar fascia from the calcaneus to the toes using maximum stretch. The other four strips of tape were attached medially and laterally to support the medial longitudinal arch with a 45° inclination. While maximum stretching was applied to the middle 1/3 of all bands, no stretching was applied to the ends. Once a week, three times
  Other Names: KinesioTex, KinesioTaping, US
  Arms: Kinesiotaping

SUMMARY:
It was aimed to compare the pain and functional results of ESWT, kinesiotherapy and corticosteroid injection in patients with treatment-resistant plantar fasciitis.

DETAILED DESCRIPTION:
The groups were randomized in patients with chronic plantar fasciitis who did not benefit from conservative treatment. A questionnaire study was conducted at the first visit, sixth week, third month, and sixth month. Visual analog scale (VAS) and The American Orthopedic Foot and Ankle Society (AOFAS) score were applied as a questionnaire at each control visit of the patients.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with PF,
* did not benefit from conservative treatment for at least six months,
* did not use anticoagulants,
* did not have bleeding disorders,
* did not have a psychiatric disease

Exclusion Criteria:

* previous ESWT or CI treatment
* obesity,
* seronegative spondyloarthropathy,
* tarsal tunnel syndrome,
* peripheral neuropathy,
* foot-ankle deformity (pes cavus, pes planus, etc.),
* history of mass around foot and ankle,
* previous foot or ankle surgery
* degenerative arthritis around this region

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain outcomes in visual analog scale (VAS) scores at six weeks in the extracorporeal shock wave therapy (ESWT) group. | Baseline and six weeks
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at week six. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain outcomes in visual analog scale (VAS) scores at three months in the extracorporeal shock wave therapy (ESWT) group | Baseline and three months
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at three months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain in visual analog scale (VAS) score at six months in the extracorporeal shock wave therapy (ESWT) group. | Baseline and six months
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at six months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain outcomes in visual analog scale (VAS) score at six weeks in the corticosteroid injection group. | Baseline and six weeks
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at six weeks. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain outcomes in visual analog scale (VAS) scores at three months in the corticosteroid injection group. | Baseline and three months
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at three months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain outcomes in visual analog scale (VAS) scores at six months in the corticosteroid injection group. | Baseline and six months
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at six months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) score at six weeks in the extracorporeal shock wave therapy (ESWT) group. | Baseline and six weeks
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at week six. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) score at three months in the extracorporeal shock wave therapy (ESWT) group. | Baseline and three months
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at three months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) score at six months in the extracorporeal shock wave therapy (ESWT) group. | Baseline and six months
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at six months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) score at six weeks in the corticosteroid injection group. | Baseline and six weeks
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at week six. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score at three months in the corticosteroid injection group. | Baseline and three months
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at three months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score at six months in the corticosteroid injection group. | Baseline and six months
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at six months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline pain in visual analog scale (VAS) score at six weeks in the kinesiotherapy group. | Baseline and six weeks
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain at week six. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain in visual analog scale (VAS) score at three months in the kinesiotherapy group. | Baseline and three months
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at three months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline pain outcomes in visual analog scale (VAS) score at six months in the kinesiotherapy group. | Baseline and six months
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at six months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) at six weeks in the kinesiotherapy group. | Baseline and six weeks
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at week six. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) at three months in the kinesiotherapy group. | Baseline and three months
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at three months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.
Change from baseline functional outcomes in the American Orthopedic Foot and Ankle Score (AOFAS) at six months in the kinesiotherapy group. | Baseline and six months
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at six months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free.

SECONDARY OUTCOMES:
Comparison of visual analog scale results of sixth-week extracorporeal shock wave therapy (ESWT), kinesiotherapy, and corticosteroid injection therapy. | sixth week
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at six months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free. We compared the VAS scores of three different treatment modalities.
Comparison of visual analog scale results of third months extracorporeal shock wave therapy (ESWT), kinesiotherapy, and corticosteroid injection therapy. | third month
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at three months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free. We compared the VAS scores of three different treatment modalities.
Comparison of visual analog scale results of sixth months extracorporeal shock wave therapy (ESWT), kinesiotherapy, and corticosteroid injection therapy. | sixth month
  The visual analog scale (VAS) score is validated, the self-reported tool that assesses the intensity of mean pain outcomes at six months. Scores range from 0 to 10; higher scores indicate greater pain intensity. The VAS score is obtained online for free. We compared the VAS scores of three different treatment modalities.
Comparison of American Orthopedic Foot and Ankle Score (AOFAS) scores results of sixth weeks extracorporeal shock wave therapy (ESWT), kinesiotherapy, and corticosteroid injection therapy. | sixth weeks
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at sixth weeks. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free. We compared the AOFAS scores of three different treatment modalities.
Comparison of American Orthopedic Foot and Ankle Score (AOFAS) scores results of three months extracorporeal shock wave therapy (ESWT), kinesiotherapy, and corticosteroid injection therapy. | three month
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at three months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free. We compared the AOFAS scores of three different treatment modalities.
Comparison of American Orthopedic Foot and Ankle Score (AOFAS) scores results of sixth months extracorporeal shock wave therapy (ESWT), kinesiotherapy, and corticosteroid injection therapy. | sixth month
  The American Orthopedic Foot and Ankle Score (AOFAS) scores are validated, self-reported tools that assess the intensity of mean functional outcomes at six months. Scores range from 0 to 100, with healthy ankles receiving 100 points. The AOFAS score is obtained online for free. We compared the AOFAS scores of three different treatment modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Orhan, Principal Investigator — Department of Orthopaedics and Traumatology, Harran University Medicine Faculty, Şanlıurfa, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Harran University Medicine Faculty, Sanliurfa, Outside of the US
  - Sanliurfa Regional Training and Research Hospital, Sanliurfa

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: for a period of six months, starting three months after publication.
Access Criteria: Information can be obtained by medical doctors by contacting the principal investigator via e-mail.

REFERENCES:
- [Result] Tang M, Wang L, You Y, Li J, Hu X. Effects of taping techniques on arch deformation in adults with pes planus: A meta-analysis. PLoS One. 2021 Jul 2;16(7):e0253567. doi: 10.1371/journal.pone.0253567. eCollection 2021. PMID 34214104
- [Result] Chang KV, Chen SY, Chen WS, Tu YK, Chien KL. Comparative effectiveness of focused shock wave therapy of different intensity levels and radial shock wave therapy for treating plantar fasciitis: a systematic review and network meta-analysis. Arch Phys Med Rehabil. 2012 Jul;93(7):1259-68. doi: 10.1016/j.apmr.2012.02.023. Epub 2012 Mar 12. PMID 22421623
- [Result] Mishra BN, Poudel RR, Banskota B, Shrestha BK, Banskota AK. Effectiveness of extra-corporeal shock wave therapy (ESWT) vs methylprednisolone injections in plantar fasciitis. J Clin Orthop Trauma. 2019 Mar-Apr;10(2):401-405. doi: 10.1016/j.jcot.2018.02.011. Epub 2018 Feb 23. PMID 30828215